CLINICAL TRIAL: NCT05468333
Title: "Natural" and "Organic" Cigarette Descriptors: Association With Expectancies, Subjective Effects, Topography, and Biomarkers of Exposure Among Daily Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Reno (Other)
Responsible Party: Principal Investigator, Jennifer Pearson, Associate Professor, University of Nevada, Reno
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5R01DA053619 (NIH)
Record Dates: First submitted 2022-07-01; First posted 2022-07-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Smoking Behaviors
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm (Experimental): All participants received the same intervention; however, the order of the intervention was randomized to reduce the risk of order effects.
  Interventions: Other: Cigarette trial

INTERVENTIONS:
Other: Cigarette trial — Participants were told that they were participating in market research for a new tobacco company called "Capital Tobacco." They were told that they were going to try three different cigarettes for the new company -- a conventional cigarette, a natural cigarette, and an organic cigarette -- and provide the research team with their impressions about the advertising and the smoking experience for each product. We also told them were were studying whether smoking these different types of cigarettes changed their exposure to chemicals in cigarette smoke. The intervention consisted of showing participants conventional, natural, and organic versions of a mailer and reading them a brief description of the brand. In reality, participants were smoking the same cigarette 3 times.

SUMMARY:
Smokers believe that cigarettes with the "natural" or "organic" descriptors are less harmful than cigarettes without these descriptors, but we do not know if these beliefs are associated with how smokers interpret the experience of smoking a "natural" or "organic" cigarette, nor whether these beliefs are predictive of changes in smoking behavior or biological exposures. The primary goal of this study is to examine the relationship between exposure to "natural" or "organic" descriptors in cigarette advertising and smoking health risk expectancies, subjective effects, topography, and biological exposures. To accomplish this goal, we will enroll 250 adult daily cigarette smokers of Natural American Spirit (NAS) or non-NAS brands (125 in each group) in a within-subjects human laboratory study manipulating four expectancy conditions (own brand comparator, "natural" advertising, "organic" advertising, "conventional" advertising).

ELIGIBILITY:
Inclusion Criteria:

* Daily cigarette smoker of 5+ cigarettes/day for at least the past 6 months and consumed 100+ lifetime cigarettes
* Smoke non-menthol, filtered cigarettes
* Report daily use of any non-Natural American Spirit (NAS) cigarette brand for the last 30 days (for the non-NAS smoker group), or report daily use of NAS cigarettes for at least 30 days (for the NAS smoker group)
* Provide exhaled CO level >= 10 ppm at the Session 1 visit
* Able to communicate fluently in English (speaking, writing, and reading)
* Capable of providing written informed consent, which includes compliance with the requirements and restrictions listed in human participant protections

Exclusion Criteria:

* Current use of Nat's cigarettes as a preferred brand
* Plan to quit smoking in the next 30 days and not currently undergoing smoking cessation treatment
* Are pregnant, planning a pregnancy, and/or lactating
* Have any impairment including, but not limited to, visual, physical, and/or neurological impairments preventing the completion of procedures included within this protocol
* Have had a serious or unstable disease within the past 6 months (e.g. heart disease, cancer, schizophrenia).
* Cannot have ever regularly smoked NAS (for the non-NAS group)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identification as a man or woman
Enrollment: 184 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Difference in perceived chemical content relative to conventional condition - natural | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  Survey measure
Difference in perceived chemical content relative to conventional condition - organic | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  Survey measure
Difference in perceived chemical aftertaste to conventional condition - natural | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  Survey measure
Difference in perceived chemical aftertaste to conventional condition - organic | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  Survey measure
Difference in total puff volume relative to conventional condition - natural | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  Total puff volume as measured by topography device
Difference in total puff volume relative to conventional condition - organic | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  Total puff volume as measured by topography device
Difference in salivary aldehyde concentration relative to conventional condition - natural | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  salivary aldehyde concentration measured in saliva
Difference in salivary aldehyde concentration relative to conventional condition - organic | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  salivary aldehyde concentration measured in saliva
Difference in perceived chemical content relative to own brand condition - natural | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  survey measure
Difference in perceived chemical content relative to own brand condition - organic | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  survey measure
Difference in perceived chemical aftertaste to own brand condition - natural | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  survey measure
Difference in perceived chemical aftertaste to own brand condition - organic | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  survey measure
Difference in total puff volume relative to own brand condition - natural | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  survey measure
Difference in total puff volume relative to own brand condition - organic | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  total puff volume as measured by a puff topography device
Difference in salivary aldehyde concentration relative to own brand condition - organic | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  salivary aldehyde concentration measured in saliva
Difference in salivary aldehyde concentration relative to own brand condition - natural | no sooner than 1 day after prior study visit and up to 3 months after first study visit.
  salivary aldehyde concentration measured in saliva

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Desert Research Institute, Reno, Nevada
  - University of Nevada, Reno, Reno, Nevada
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT05468333/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT05468333/ICF_001.pdf